CLINICAL TRIAL: NCT07124442
Title: Relationship of Disease Severity and Mortality Risk With Respiratory Muscle Strength, Muscle Biomechanical Properties, and Muscle Architecture in Intensive Care Unit Patients
Brief Title: Disease Severity, Mortality Risk, and Muscle Function in Intensive Care Unit Patients
Status: Recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Beyza Tanrıöğen, Research Assistant (PhD student), Istinye University
Other Study IDs: Istinye BT 2
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Critically Ill Patients
Keywords: Critically ill patients; Respiratory muscle; Skeletal muscle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical care patient: Critical care patients are going to be meaasured

SUMMARY:
Intensive Care Units are specialized, technologically advanced hospital units that provide continuous monitoring and care from multiple healthcare disciplines for patients who are critically ill and face a high risk of death or serious health problems. Prolonged periods of immobility, which are common during treatment in these units, can cause serious complications such as muscle weakness, decline in physical function, and a lower quality of life. There are scoring systems designed to predict the severity of a patient's illness and their likely outcomes, such as the scoring system called the Acute Physiology and Chronic Health Evaluation version two. However, these scoring systems are not yet widely used as a regular part of patient care. Although weakness and wasting of muscles away from the center of the body are known to affect the recovery process of patients who survive intensive care treatment, the connection between how severe the illness is and the strength of the muscles used for breathing, the structure of peripheral muscles, and their biomechanical characteristics is still not fully understood. This study aims to explore these relationships to help improve physiotherapy and rehabilitation treatments for patients in intensive care.

DETAILED DESCRIPTION:
Intensive Care Units are specialized and high-cost hospital units equipped with advanced technology, designed for the treatment and continuous monitoring of critically ill patients who are at risk of losing, or have already lost, some or all of their vital bodily functions. These units provide twenty-four-hour monitoring of vital signs, operate with a multidisciplinary healthcare team, and have privileged status in terms of patient care (1). The most common reasons for admission to Intensive Care Units include acute heart attacks, severe breathing difficulties, heart bypass surgeries, congestive heart failure, strokes or bleeding within the brain, cardiovascular system problems, pneumonia, widespread infections called sepsis, diabetic ketoacidosis, gastrointestinal bleeding, and other serious health conditions (2). Among these, the most frequent reason for admission is respiratory failure that requires mechanical support to assist or take over breathing (3). The period of critical illness can last from a few hours to several months depending on the underlying disease process and how the patient responds to treatment, and it is associated with high rates of death and serious health problems (4).

Patients treated in Intensive Care Units face various problems that either develop during their stay or exist beforehand and continue. These problems include muscle weakness, cognitive difficulties, psychological challenges, worsening physical function, and reductions in quality of life and the ability to perform daily activities (5). Bed rest or immobilization is often a necessary part of treatment in Intensive Care Units (3). Prolonged immobility can cause many clinical complications that may be severe and last a long time, leading to physical limitations and negatively affecting quality of life over the long term (6). Research has identified bed rest as harmful because it can cause complications such as fluid buildup in the lungs, collapse of parts of the lungs, loss of bone density, muscle wasting, instability of blood vessel regulation, constipation, pain, pressure sores, joint contractures, and blood clots (7).

Predictive scoring systems are clinical tools used to evaluate the severity of illness in Intensive Care Unit patients and to predict their prognosis, especially the risk of death (8). These clinical scoring systems help classify patient risk levels, predict health outcomes, and improve other clinical management processes. Although these scoring tools assist physicians in managing patients, they are not routinely used in everyday clinical practice mainly because they are complex and require specific expertise and training (9).

Some of the common scoring systems used for adult patients in Intensive Care Units include the Acute Physiology and Chronic Health Evaluation, the Simplified Acute Physiology Score, the Mortality Prediction Model, the Organ Dysfunction and Infection System, the Sequential Organ Failure Assessment, the Multiple Organ Dysfunction Score, the Logistic Organ Dysfunction Model, and the Three-day Recalibrating Intensive Care Unit Outcomes system (10).

The Acute Physiology and Chronic Health Evaluation scoring system was developed in nineteen eighty-one by the George Washington University Medical Center and is known as one of the most widely used and recognized scales for determining the severity of acute illnesses. The version known as Acute Physiology and Chronic Health Evaluation version two was created for different research and clinical audit purposes and continues to be used extensively to assess disease severity in critically ill patients in Intensive Care Units (11, 12). It is a highly selective and accurate measurement tool that can serve as a standard in Intensive Care Units by enabling evaluation of standardized mortality ratios (12).

Loss of muscle strength and muscle weakness are well known to negatively impact patients in Intensive Care Units. This loss of muscle strength can delay or hinder the recovery of physical function in patients who survive Intensive Care Unit treatment. Additionally, patients who develop muscle weakness due to long stays in Intensive Care Units have been shown by ultrasound measurements to have reduced thickness and cross-sectional area of peripheral muscles compared to patients without muscle weakness (13, 14). However, the relationship between the course and severity of disease and respiratory muscle strength, peripheral muscle thickness, and muscle tone in Intensive Care Unit patients is not yet fully understood. Determining how the course and severity of disease affect respiratory muscle strength, biomechanical properties of peripheral muscles, and muscle structure is critically important for establishing effective physiotherapy and rehabilitation strategies in Intensive Care Units.

The aim of this study is to investigate the relationship between disease severity and respiratory muscle strength, peripheral muscle structure, and the biomechanical properties of peripheral muscles in patients treated in Intensive Care Units. This study will be conducted using a cross-sectional and observational research design.

ELIGIBILITY:
Inclusion Criteria:

Not dependent on mechanical ventilation,

Patient or legal representative provides consent to participate,

Aged 18 years or older,

Monitored in the ICU for at least 48 hours.

Exclusion Criteria:

Unable to obtain ethical consent,

Presence of neuromuscular disease affecting muscle tone,

Patients unable to cooperate during measurement due to impaired consciousness, communication disorder, or other medical reasons,

Presence of infection, open wound, or any lesion impairing skin integrity at the anatomical measurement site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit who are not dependent on mechanical ventilation and meet the inclusion and exclusion criteria will be included in the study.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Course of Disease in Intensive Care Patients, Mortality risk: | 4 weeks
  The patient's mortality rate will be assessed using the Acute Physiology and Chronic Health Evaluation II score. The Acute Physiology and Chronic Health Evaluation II score is commonly used for patients treated in the intensive care unit. It is based on an initial score comprising 12 components and is evaluated on a scale from 0 to 71 points. The assessment consists of three sections: physiological scores ranging from 0-60 points, age scores ranging from 0-6 points, and comorbidity scores ranging from 0-5 points. A higher total Acute Physiology and Chronic Health Evaluation II score indicates greater severity of the patient's condition (15).
Assessment of Peripheral Muscle Architecture: | 4 weeks
  Quadriceps femoris muscle thickness will be measured as the distance between the upper border of the femur and the lower border of the subcutaneous tissue. Measurements will be taken 15 cm proximal to the superior border of the patella using a tape measure (19). After each patient, the ultrasound probe will be disinfected by wiping with 70% isopropyl alcohol.

SECONDARY OUTCOMES:
Muscle Tone: | 4 weeks
  Peripheral muscle stiffness will be assessed using the MyotonPRO device (Myoton AS, Estonia). Tone refers to the tension of the tissue at rest. There is a direct relationship between the measured value and tissue tension.
Measurement of Respiratory Muscle Strength: | 4 weeks
  Respiratory muscle strength will be assessed using a portable electronic device (Micro Medical Micro RPM, Rochester, UK) to measure maximal inspiratory mouth pressure and maximal expiratory mouth pressure in cmH₂O. Maximal inspiratory mouth pressure is recorded during maximal inspiration against an occluded airway after full expiration, sustained for 1-3 seconds; maximal expiratory mouth pressure is recorded during maximal expiration after full inspiration. The best of three trials will be expressed as a percentage of age- and sex-adjusted reference values. To prevent infection, disposable mouthpieces and filters will be used, with device surfaces disinfected using alcohol-based solutions, and mouthpieces sterilized with ethyl alcohol and specialized equipment.
Elasticity: | 4 weeks
  It will be measured by using the MyotonPRO device (Myoton AS, Estonia). Elasticity is the ability of the tissue to return to its original shape after the removal of deforming forces. Tissue elasticity and the measured value are inversely related; as the logarithmic decrement decreases, the tissue's ability to return to its original shape increases.
Dynamic Stiffness | 4 weeks
  Peripheral muscle stiffness will be assessed using the MyotonPRO device (Myoton AS, Estonia). Dynamic stiffness (measured in Newtons per meter, N/m) is defined as the resistance of soft tissues to destructive external forces. Tissue stiffness and the measured value are inversely related.
Creep: | 4 weeks
  Peripheral muscle stiffness will be assessed using the MyotonPRO device (Myoton AS, Estonia). Creep is the gradual elongation of soft tissue over time under a constant load. It is calculated as the ratio of deformation time to tissue relaxation time. Higher values are typically found in young, healthy muscles.
Relaxation Time: | 4 weeks
  Peripheral muscle stiffness will be assessed using the MyotonPRO device (Myoton AS, Estonia). Relaxation time (measured in milliseconds) is the time required for tissue to recover after deformation or damage. There is a direct relationship between the measured value and the time taken for full recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University Bahçeşehir Liv University Hospital, Istanbul, Esenyurt, Turkey (Türkiye)